CLINICAL TRIAL: NCT04825106
Title: Context-dependent Diagnostic Accuracy in Anaphylactic Shock
Brief Title: Diagnostic Errors in Anaphylactic Shock
Acronym: ANASim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 4031-Sim-ANA
Record Dates: First submitted 2021-03-22; First posted 2021-04-01 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Diagnostic Error

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Expected (Active Comparator): Anaphylactic shock occurs after the injection of a drug known to cause allergic reactions
  Interventions: Other: Diagnostic context
- Unexpected, no distractor (Active Comparator): Anaphylactic shock occurs unexpectedly, but their is no medical distractor
  Interventions: Other: Diagnostic context
- Unexpected, with distractor (Active Comparator): Anaphylactic shock occurs unexpectedly. Scenario is set up such, that a tension pneumothorax may be a likely explanation
  Interventions: Other: Diagnostic context

INTERVENTIONS:
Other: Diagnostic context — A life-threatening situation occurs in 3 different contexts

SUMMARY:
Diagnostic accuracy and quality of management in anaphylactic shock is assessed in three conditions: expected, unexpected with no distractor, unexpected with distractor

DETAILED DESCRIPTION:
participants: physicians taking part in voluntary workshops. Participants are allocated to teams of three design: prospective, randomized, single-blind setting: simulated anaphylactic shock intervention: participants are allocated to 3 versions of the scenario: 1) expected, 2) unexpected but no distractor, 3) unexpected with distractor

ELIGIBILITY:
Inclusion Criteria:

* Physicians taking part in voluntary simulator workshops

Exclusion Criteria:

* Refusal to participate or to being videorecorded

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Correct diagnosis of anaphylactic shock | 15 minutes
  Diagnosis of anaphylactic shock is explicitly stated by at least one team member within a time frame of 15 minutes after onset

SECONDARY OUTCOMES:
Treatment of anaphylactic shock with epinephrine ≥ 0.3mg intravenously | 5 minutes
  Anaphylactic shock is correctly treated with epinephrine in an appropriate dose (≥ 0.3mg intravenously) within a time frame of 5 minutes after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Marsch, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No
Secondary data can be shared Videorecordings are strictly confidential and cannot be shared